CLINICAL TRIAL: NCT03664141
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Pilot Study to Investigate the Safety and Efficacy of Cannabis Oil in Maintenance Hemodialysis Patients With Protein-energy Wasting
Brief Title: Impact of Cannabis Oil on Nutrition in Hemodialysis Patients Study (ICON-HP Study)
Acronym: ICON-HP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: TIKUN OLAM has not received approval from the National Committee to conduct research
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Tikun Olam (Unknown)
Responsible Party: Principal Investigator, ilia beberashvili MD, principal investigator, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Assaf Harofeh MC
Record Dates: First submitted 2018-07-20; First posted 2018-09-10 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2018-09

CONDITIONS: Protein-Energy Malnutrition; Hemodialysis; Appetite Disorders
Keywords: Malnutrition; Hemodialysis; Appetite; Inflammation; Body composition; Cannabis oil
MeSH Terms: conditions — Protein-Energy Malnutrition; Feeding and Eating Disorders; Malnutrition; Inflammation | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): 1 drop of regular oil for food labeled as 3% cannabis oil once a day during 3 months
  Interventions: Drug: Cannabis oil; Drug: Placebo/ Regular Oil
- Cannabis oil group (Experimental): 1 drop of 3% cannabis oil once a day during 3 months
  Interventions: Drug: Cannabis oil; Drug: Placebo/ Regular Oil

INTERVENTIONS:
Drug: Cannabis oil — Treatment with cannabis oil
Drug: Placebo/ Regular Oil — Treatment with placebo (Regular Oil)

SUMMARY:
The study will be performed in two parts: 1) The pharmacokinetic (PK) part and 2) The appetite and nutritional evaluation part.

The PK part of study will be conducted in open label manner on 10 end stage kidney disease (ESKD) patients receiving maintenance hemodialysis (MHD) treatment. For the PK part, a starting dose of cannabis oil -1 drop of 3% cannabis oil once a day [each drop contain 1.2 mg CBD (cannabidiol) and 1.2 mg of ∆9-THC (∆9-tetrahydrocannabinol)], was judged to be safe for a first-in-MHD patient's administration. Escalation to the next higher dose and any dose adjustments of the next dose levels will be based on safety and tolerability results of the previously administered dose and available PK data of previous dose groups. Once the first dosage proved to be safe, there will be a 2 fold increase from the first dose level (2 drops once a day) to the second dose level. The dose levels will be increased by 2-fold from the previous dose level, until basal hunger and prospective consumption ratings assessed by the visual analogue scale (VAS) will increase at least by 10 mm between screening and the study visits (change-from-baseline) . PK parameters will be evaluated after first dosage administration and after dosage increased.

The appetite and nutritional evaluation part of study will be conducted as a 3-month, double-blind, parallel-group, placebo-controlled, single center study. The study population will include 30 ESKD patients receiving MHD treatment with different degrees of protein-energy wasting (PEW) defined as malnutrition-inflammation score (MIS) above 6. A total of 30 subjects will be randomized to treatment with either cannabis oil or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age > 18 years, on MHD hemodialysis treatment at least 3 months
* Stable and adequate hemodialysis treatment three months prior to participation in study as defined by Kt/V > 1.2 and/or hemodialysis performed 4 hours 3 times weekly
* Patients with Malnutrition-Inflammation Score (MIS) ≥ 6
* Informed consent obtained before any trial-related activities

Exclusion Criteria:

* Previous or current use in cannabis or marijuana
* Critical illness as defined by the need of respiratory or circulatory support
* Known or suspected allergy to trial products
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using contraceptive methods
* Patients with active malignant disease or liver cirrhosis
* Actively symptomatic gastrointestinal bleeding and inflammatory bowel disease
* Patients on chronic treatment with steroids on doses > 10 mg/day Prednisone (or equivalent)
* Patients treated with immunosuppressive agents
* Patients receiving any of the following medications: Astemizole, Cisapride, Pimozide or Terfenadine
* Patients suffering from:

  * Acute vasculitis
  * Severe systemic infections
  * Severe Heart failure (NYHA class IV)
  * Severe hepatic disease, defined as ALT or AST levels >3 times upper normal range
  * Mental incapacity, unwillingness or language barrier
* Any condition judged by the investigator to interfere with trial participation or evaluation of results or to be potentially hazardous to the patient
* A significant history of alcohol, drug or solvent abuse
* History of schizophrenia, affective disorder, history of psychiatric hospitalization and diagnosed anxiety disorder
* The receipt of any investigational drug within 1 month prior to initiating of this study
* Scheduled renal transplantation (fixed date).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2019-08-15 (Estimated); Study Completion 2019-10-15 (Estimated)

PRIMARY OUTCOMES:
Overall incidence and prevalence of adverse events | For 5 months from the day of randomization
  Overall incidence and prevalence of adverse events
Change in appetite assessed by the Visual Analogue Scale (VAS). | For 5 months from the day of randomization
  VAS, 100 mm in length with words anchored at each end, expressing the most positive (=100) and the most negative rating (=0), will be used to assess specific domains of appetite separately: hunger, satiety, fullness, prospective food consumption. Each domain will be measured by the 0-100mm scale as mentioned above.

SECONDARY OUTCOMES:
Change in nutritional status assessed by the Malnutrition-Inflammation Score (MIS). | For 5 months from the day of randomization
  MIS consists of four sections (nutritional history, physical examination, body mass index [BMI], and laboratory values) and 10 components. Each MIS component has four levels of severity from 0 (normal) to 3 (very severe). The sum of all 10 components results in an overall score ranging from 0 (normal) to 30 (severely malnourished).
Change in Health Related Quality of Life assessed by short form 36 (SF-36) quality of life (QoL) scoring system | For 5 months from the day of randomization
  SF-36 consists of 36 questions, 35 of which are compressed into eight multi-item scales:
  (1) physical functioning; (2) role-physical (3) bodily pain ; (4) general health; (5) vitality ; (6) social functioning (7) role-emotional and (8) mental health. In the SF36 scoring system, the scales are assessed quantitatively, each on the basis of answers to two to ten multiple choice questions, and a score between 0 and 100 is then calculated on the basis of well-defined guidelines, with a higher score indicating a better state of health.

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf ha Rofeh, MC, Zrifin, Israel

IPD SHARING:
Plan to Share IPD: No